CLINICAL TRIAL: NCT03960515
Title: Cardiovascular Risk, Myocardial Fibrosis and Heart Failure in Rheumatoid Arthritis: Screening and Prognosis
Brief Title: Cardiovascular Profiles in Rheumatoid Arthritis
Acronym: RA-HF
Status: Completed | Type: Observational
Sponsor: Maria Betânia Almeida Dias Ferreira (Other)
Collaborators: Instituto de Ciências Biomédicas Abel Salazar (Other); Central Hospital, Nancy, France (Other); Unit Multidisciplinary Research in Biomedicine (Unknown)
Responsible Party: Sponsor-Investigator, Maria Betânia Almeida Dias Ferreira, Internal Medicine Medical Doctor, PhD student, Centro Hospitalar do Porto
Organization: Centro Hospitalar do Porto (Other)
Other Study IDs: 2016-023 (020-DEFI/020-CES)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure; Cardiovascular Risk Factor; Rheumatoid Arthritis; Myocardium; Injury; Cardiovascular Diseases
Keywords: Rheumatoid Arthritis; Heart disease; Cardiovascular Risk
MeSH Terms: conditions — Heart Failure; Arthritis, Rheumatoid; Wounds and Injuries; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease is the leading cause of death in RA patients. This increased risk may be apparent even before the clinical recognition of RA. The optimal approach for identification of patients with increased CV risk has yet to be fully established and a substantial proportion of RA patients at high risk remain unidentified.

Heart failure (HF) has been recently recognized as an important contributory factor to the excess CV mortality associated with RA (more than myocardial ischemia), and RA patients with concomitant HF have twice the risk of CV death compared with patients with RA alone. HF in RA typically presents with occult or atypical clinical symptomatology, tend to be managed less aggressively and have poorer outcomes.

For developing effective preventive strategies, the evaluation of patients in early asymptomatic stages is of great importance.

The investigators propose to perform an observational longitudinal study (with cases and controls) including RA patients (with and without HF) from a single centre to determine cardiovascular profiles that may be associated with higher risk for developing symptomatic HF and CV events. For this purpose the investigators will use clinical, echocardiographic, serum biomarker, and genetic data

DETAILED DESCRIPTION:
Patient Selection:

Screen ~400 Rheumatoid Arthritis (RA) patients followed in Centro Hospitalar do Porto outpatient clinic. All RA patients with regular follow-up will be potentially included.

The investigators also aim to enrol age-matched controls for biomarker comparison.

Experimental Design:

Observacional study with matched control. No intervention will be performed. Outpatients fulfilling the inclusion criteria will be invited to participate in the study. All patients will have to sign written informed consent to participate in the study.

An external and independent data verification will be performed. The total trial enrolment period was 23 months. . Participants will continue to receive treatments as clinically indicated and according to the decision of their attending physicians.

A structured evaluation will be performed. Every 4 to 6 months the participants will be observed in the clinic for their physicians according clinic protocol. The participants will not require additional visits to the hospital other than the visits already prespecified by their attending physicians.

Clinical Evaluation:The clinical evaluation will be performed to all RA patients and for age-matched controls Each participant and group control will be evaluated for their cardiovascular symptoms, history and risk factors for cardiovascular disease, other comorbiditys as renal disease, dementia, liver or respiratory disease or anemia. The participants will be evaluated for their Rheumathoid Arthritis history (diagnosis date, rx erosion, other autoimune diseases or treatment). All will perform a 6-minute walk test (6MWT), point blood pressure, heart rate, chest exam, ankle-brachial index, measurement of abdominal circumference and visceral fat, disease activity score 28 (DAS-28), quality of life scores (QoL), Graffar scale (socio-economic), Mini-cog and Epworth scale.

Cardiac Function: Each participant will undergo a 12 lead ECG and a transthoracic echocardiography. M-mode, 2D and Doppler measurements will be acquired according to standard recommendations. LV mass and LV mass index, left atrial (LA) volume, LA volume index, isovolumetric relaxation time (IVRT), mitral inflow E to A ratio (mitral E/A), mitral deceleration time of early filling (mitral DT), PW Doppler early diastolic velocity of the septal (septal e') and lateral (lateral e') mitral annulus, mitral inflow E velocity to early diastolic tissue Doppler of both the septal (septal E/e') and lateral (lateral E/e') mitral annulus and the pulmonary artery systolic pressure (PASP) will be measured using standard techniques19. All measurements reflect an average of at least 4 consecutive cardiac cycles and will be performed by an experienced echocardiographer.

Regular Plasma and Urine Biomarkers:For all participants. Regular blood biomarkers: hemoglobin, hematocrit, RDW, Thrombocytes, Leucocytes, lymphocytes, neutrophils, NT-proBNP , Troponin I, C-reactive Protein, Alkaline phosphatase, Ƴ-GT, Sedimentation rate, Glucose, Total Cholesterol, Triglycerides, LDL-Cholesterol,HDL- Cholesterol, Transferrin saturation, Ferritin, HbA1c, Pre-albumin, C-Cistatin, homocystein, Sodium , Potassium, Chlorine, Calcium, Phosphorus, Magnesium, Creatinine, Urea, Folic Acid, Cianocobalamin, PTH, eGFR, D Vitamin, Uric Acid.

Urine biomarkers: Microalbumin, Creatinine, Potassium, Sodium.

Specific biomarkers: For all RA patients and control group. Include OLINK's panels for inflammation, fibrosis or matrix extracellular organization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid arthritis
* Regular follow up on Autoimmune diseases medical appointment
* Written informed consent to participate in this study prior to any study procedures

Exclusion Criteria:

* Presence of severe life-threatening disease before inclusion with an expected survival of less than 6 months after inclusion
* Mental or physical status not allowing written informed consent
* Active malignancy disease
* Patient unable to walk, in which SMWT is not possible to perform.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with diagnosis of Rheumatoid Arthritis.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Number of dead participants | 11 to 32 months
  Death of any cause
Number of Participants with New diagnosis of heart failure | 11 to 32 months
  New onset of heart failure symptons with diuretic drugs starting

SECONDARY OUTCOMES:
Number of Participants with worsening of previous heart failure | 11 to 32 months
  Worsening of heart failure with increase of diuretic or diuretic IV
Number of Participants with new onset atrial fibrillation | 11 to 32 months
  New onset of Atrial Fibrillation
Number of Participants with Hospitalization | 11 to 32 months
  Any hospitalization for urgent or unplanned reasons
Number of Participants with new onset of stroke or Transient ischemic attack | 11 to 32 months
  New onset of stroke or transient ischemic attack
Number of Participants with New onset of acute myocardial infarction | 11-32 months
  New onset of acute myocardial infarction?

CONTACTS AND LOCATIONS:
Overall Officials: António J. Marinho, MD, PhD, Study Chair — Centro Hospitalar do Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibofsky A. Overview of epidemiology, pathophysiology, and diagnosis of rheumatoid arthritis. Am J Manag Care. 2012 Dec;18(13 Suppl):S295-302. PMID 23327517
- [Background] Choy E, Ganeshalingam K, Semb AG, Szekanecz Z, Nurmohamed M. Cardiovascular risk in rheumatoid arthritis: recent advances in the understanding of the pivotal role of inflammation, risk predictors and the impact of treatment. Rheumatology (Oxford). 2014 Dec;53(12):2143-54. doi: 10.1093/rheumatology/keu224. Epub 2014 Jun 6. PMID 24907149
- [Background] Kawai VK, Chung CP, Solus JF, Oeser A, Raggi P, Stein CM. The ability of the 2013 American College of Cardiology/American Heart Association cardiovascular risk score to identify rheumatoid arthritis patients with high coronary artery calcification scores. Arthritis Rheumatol. 2015 Feb;67(2):381-5. doi: 10.1002/art.38944. PMID 25371313
- [Background] Agca R, Heslinga SC, Rollefstad S, Heslinga M, McInnes IB, Peters MJ, Kvien TK, Dougados M, Radner H, Atzeni F, Primdahl J, Sodergren A, Wallberg Jonsson S, van Rompay J, Zabalan C, Pedersen TR, Jacobsson L, de Vlam K, Gonzalez-Gay MA, Semb AG, Kitas GD, Smulders YM, Szekanecz Z, Sattar N, Symmons DP, Nurmohamed MT. EULAR recommendations for cardiovascular disease risk management in patients with rheumatoid arthritis and other forms of inflammatory joint disorders: 2015/2016 update. Ann Rheum Dis. 2017 Jan;76(1):17-28. doi: 10.1136/annrheumdis-2016-209775. Epub 2016 Oct 3. PMID 27697765
- [Background] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Background] Arts EE, Popa C, Den Broeder AA, Semb AG, Toms T, Kitas GD, van Riel PL, Fransen J. Performance of four current risk algorithms in predicting cardiovascular events in patients with early rheumatoid arthritis. Ann Rheum Dis. 2015 Apr;74(4):668-74. doi: 10.1136/annrheumdis-2013-204024. Epub 2014 Jan 3. PMID 24389293
- [Derived] Ferreira MB, Fonseca T, Costa R, Marinho A, Oliveira JC, Zannad F, Rossignol P, Rodrigues P, Barros AS, Ferreira JP. Sex differences in circulating proteins of patients with rheumatoid arthritis: A cohort study. Int J Rheum Dis. 2022 Jun;25(6):669-677. doi: 10.1111/1756-185X.14323. Epub 2022 Apr 15. PMID 35429115
- [Derived] Ferreira MB, Fonseca T, Costa R, Marinhoc A, Carvalho HC, Oliveira JC, Zannad F, Rossignol P, Gottenberg JE, Saraiva FA, Rodrigues P, Barros AS, Ferreira JP. Prevalence, risk factors and proteomic bioprofiles associated with heart failure in rheumatoid arthritis: The RA-HF study. Eur J Intern Med. 2021 Mar;85:41-49. doi: 10.1016/j.ejim.2020.11.002. Epub 2020 Nov 6. PMID 33162300